CLINICAL TRIAL: NCT03808129
Title: The Evaluation of Ultrasonography-guided Erector Spinae Plane Block in Perioperative Analgesia and Intraabdominal Tissue Oxygenation in Pediatric Patients Undergoing Lower Abdominal Surgery
Brief Title: Erector Spinae Plane Block for Peroperative Analgesia and Intraabdominal Tissue Oxygenation
Acronym: ESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P0001
Record Dates: First submitted 2018-12-13; First posted 2019-01-17 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Lower Abdominal Surgery
Keywords: erector spinae plane block; postoperative analgesia; RSO2
MeSH Terms: interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: As the patients were under 18 years of age, the details of the procedure were explained to their parents and their consent was obtained. However, the patients were not included in the group. And also outcomes assessor staff were not aware of medication assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group: Bupivacaine and lidocaine (Active Comparator): ESP Group: Bupivacaine and lidocaine: Erector Spinae Plane Block : (1: 1 ratio of 0.25% bupivacaine and 0.4 ml / kg of 1% lidocaine) was administered.
  Interventions: Drug: Bupivacaine and Lidocaine
- control group (No Intervention): Control Group:

INTERVENTIONS:
Drug: Bupivacaine and Lidocaine — ESP block was administered under general anesthesia before the surgery. Patients with ESP block, 1: 1 ratio of 0.25% bupivacaine and 0.4 ml / kg of 1% lidocaine
  Other Names: ESP block
  Arms: ESP Group: Bupivacaine and lidocaine

SUMMARY:
Brief summary: Regional anesthesia decreases the need for intravenous analgesia in the peri-operative period. Erector spinae plane (ESP) is a regional anesthesia technique shown to be effective at the dorsal and ventral rami of the thoracic spinal nerve along with sympathetic nerve fibers. The purpose is to demonstrate the contribution of ESP block to the postoperative analgesia by ultrasonography and to increase intraabdominal tissue oxygenation compared to the control group.

DETAILED DESCRIPTION:
50 patients with American Society of Anesthesiologists (ASA) physical score I-II were randomly divided into 25 patients in the ESP group and 25 patients in the control group. Patients were premedicated with oral midazolam 0.5 mg kg-1, 30 minutes before surgery Anesthesia monitorization was made with electrocardiogram, non-invasive blood pressure, peripheral oxygen saturation (SpO2), end-tidal carbon dioxide, temperature, Bispectral index (BIS), and Regional tissue saturation (rSO2). Anesthesia was induced with a face mask distributing 8% sevoflurane and 50% air in oxygen while the patients were breathing spontaneously. After anesthesia induction, peripheral venous access was established and propofol 2 mg kg-1 and fentanyl citrate 1 μg kg-1 were administered. Laryngeal mask airways were used to secure the upper airways. Anesthesia was maintained with sevoflurane and 50% air in oxygen. The concentration of sevoflurane was adjusted by targeting BIS scores at 50-60 in all groups. During the operations, fentanyl was administered at a dose of 0.5 μg kg-1 if the blood pressure and heart rates were 20% higher than the baseline value. In ESP blok groups, after general anesthesia induced, patients were placed in the lateral position and ESP block was performed under ultrasound guidance. For ESP block, 1: 1 ratio of 0.25% bupivacaine and 0.4 ml / kg of 1% lidocaine was administered. In all groups, regional tissue saturation (RSO2) was evaluated Continuously with near infrared spectroscopy (NIRS) probe from anesthesia induction to the end of surgery. Commercially available device (INVOS Cerebral Oximeter; somatics Corp, Troy, Mich) was used to monitor rSO2 values in the surgery side flank during surgical intervention. Pain was evaluated and recorded using the FLACC (Face, Legs, Activity, Cry, Consolability) scale at the 1st, 2nd, 8th, 12th and 24th hours. Total analgesic consumption was recorded during the operation and postoperative time to first analgesic drug and number of patients who required analgesic in the first 24 hours, parents satisfaction score, discharge time as well as adverse effects such as nausea and vomiting were recorded in the postoperative periods.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 months to 2 years
2. According to American Anesthesia Society Anesthesia Risk Scale ASA I-II class patients
3. Patients with lower abdominal surgery

Exclusion Criteria:

1. Children under 6 months and older than 2 years
2. According to American Anesthesia Society Anesthesia Risk Scale Patients with ASA III-IV class
3. Patients with contraindication to regional anesthesia
4. Patients with a history of local anesthetic allergy
5. Patients with abnormal coagulation profile
6. Patients with infection at the injection site

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
FLACC scale | From recovery of anesthesia to end of study ( postoperative 24 hours)
  FLACC scale was used. The Face, Legs, Activity, Cry, Consolability scale (FLACC) scale was a measurement used to assess pain for children between the ages of 6 months and 2 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
NIRS | Before anesthesia induction to end of operation ( intraoperative 2 hours )
  INVOS ;Somatic Corp, Troy, Mic sensors placed in surgical side of patients was used to detect peripheral perfusion and oxygen delivery (rSo2)

SECONDARY OUTCOMES:
Time to first analgesic drug | first 24 hour
  Time to first analgesic drug will be recorded
Need for analgesic | first 24 hour
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: PARVIN PINAR, Study Chair — BEZMİALEM VAKIF UNIVERSITY
Locations (1):
- Parvin Pinar, Istanbul, Turkey (Türkiye)